CLINICAL TRIAL: NCT00754377
Title: Developing a PBLI QI Systems Impact Assessment Questionnaire
Brief Title: Developing a Practice-Based Learning and Improvement Quality Improvement (QI) Systems Impact Assessment Questionnaire
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SHP 08-194
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Quality Improvement
Keywords: Education; Program Evaluation; Quality of Health Care; Medical Residents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PBLI Curriculum group: To evaluate preliminary data on a PBLI curriculum grounded on QI system projects.
  Interventions: Other: PBLI Curriculum
- Comparison group: Received a different curriculum.

INTERVENTIONS:
Other: PBLI Curriculum — PBLI curriculum was offered on alternate rotations
  Groups: PBLI Curriculum group

SUMMARY:
The Accreditation Council for Graduate Medical Education (ACGME) acknowledged the changing needs of physicians in training when it endorsed practice-based learning and improvement (PBLI) -- a competency that is typically omitted from medical curriculum. The goal is to have residents competent to investigate and evaluate their own patient care practices, integrate scientific evidence and be able to improve their practices. Available assessment tools do not adequately address all of the components of PBLI and few assessment tools attempt to capture the residents' ability to develop and implement clinically-based Continuous Quality Improvement (CQI) projects that involve the practice setting. Curriculums without such foci miss the importance of system perspectives and opportunities for interprofessional team development. Our aim is to evaluate preliminary data on the curriculum we developed to address the gaps, to develop an assessment tool, and to provide methods for assessing the sustainability of system projects.

The key component of the curriculum is the integration of system quality improvement projects. PBLI curriculum was offered on alternate rotations. Preliminary data is available from 6 PBLI QI Systems Curriculum blocks (n=50) and 5 comparison blocks (n=42). Data includes closed- and open-ended questions designed to assess resident PBLI application skills, the notes and presentation slides for the residents' presentation.

DETAILED DESCRIPTION:
Physicians in training operate in complex healthcare delivery systems but many have not been equipped with the knowledge or skills to analyze clinical environments and continually improve patient care.[1] Instead, their training emphasizes the clinical management of individual patients. The Accreditation Council for Graduate Medical Education (ACGME) acknowledged the changing needs of physicians in training when it endorsed one of two novel core competencies that are typically omitted from formal medical curriculum: practice-based learning and improvement (PBLI).[2,3] The ACGME's PBLI competency involves six points. The overall objective is to have residents competent to investigate and evaluate their own patient care practices, evaluate and integrate scientific evidence into their clinics and be able to improve their practices. However, the ACGME was not prescriptive about how to successfully implement and evaluate PBLI, and an established curriculum and validated assessment tool did not exist.[4] Efforts to date to develop an assessment tool provide a foundation, but none adequately addresses all of the components of PBLI as described by the ACGME. [3, 5-10] In particular, few assessment tools attempt to capture the residents' ability to develop and implement clinically-based CQI projects that involve the practice setting and assess impact on the practice setting and/or organization. Curriculums without such foci miss the importance of system perspectives, opportunities for interprofessional team development, and meaningful impacts on patient care at a broader organizational level.

After several iterations, a PBLI QI curriculum that addressed the gaps identified in many other curriculums was instituted. [11] The key component was the integration of system quality improvement projects that could evolve over several resident outpatient rotation blocks. Data from 11 blocks of the new curriculum is available for analysis. Data includes closed- and open-ended questions designed to assess resident PBLI application skills and the notes and presentation slides for the residents' presentation at the internal medicine's morbidity and mortality conference (IM MMC) at the end of each block. Funding would make it possible to more quickly evaluate the existing preliminary data. Our overall aim is to evaluate the preliminary data on the new curriculum and develop an assessment tool that addresses the six ACGME points and provides methods for assessing the sustainability of system projects. The next step will be to apply for a grant to more fully evaluate the curriculum and assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* None, data being used has already been collected from a previous study which the inclusion criteria included all Internal Medicine and Medicine-Pediatrics residents completing a 4 week ambulatory block from 2005-2006 were required to participate in the PBLI curriculum to satisfy an ACGME's core competency.

Exclusion Criteria:

* None, the residents from 2004 that did not complete a 4 week ambulatory block and residents participating in ambulatory block 7 and 13 were excluded from the study previously Institutional Review Board (IRB) approved and exempted study. Blocks 7 and 13 are not structured to permit teaching.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Internal Medicine residents
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Aron, MD MS, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

REFERENCES:
- [Result] Stulberg JJ, Delaney CP, Neuhauser DV, Aron DC, Fu P, Koroukian SM. Adherence to surgical care improvement project measures and the association with postoperative infections. JAMA. 2010 Jun 23;303(24):2479-85. doi: 10.1001/jama.2010.841. PMID 20571014
- [Result] Lawrence RH, Tomolo AM. Development and preliminary evaluation of a practice-based learning and improvement tool for assessing resident competence and guiding curriculum development. J Grad Med Educ. 2011 Mar;3(1):41-8. doi: 10.4300/JGME-D-10-00102.1. PMID 22379522
- [Result] Tomolo AM, Lawrence RH, Watts B, Augustine S, Aron DC, Singh MK. Pilot study evaluating a practice-based learning and improvement curriculum focusing on the development of system-level quality improvement skills. J Grad Med Educ. 2011 Mar;3(1):49-58. doi: 10.4300/JGME-D-10-00104.1. PMID 22379523

RESULTS

PARTICIPANT FLOW:
Groups:
- PBL Curriculum Group: To evaluate preliminary data on a PBLI curriculum grounded on QI system projects.
  PBLI curriculum comparison: The design is a pre-post comparison of PBLI curriculum participants versus non-participants. Data will come from the closed-ended items on the questionnaire given before the rotation and at the end of the rotation. PBLI curriculum was offered on alternate rotations (residents on alternate month were involved with a different curriculum). Preliminary data is available from 11 blocks, 6 PBLI QI Systems Curriculum blocks (n=50) and 5 comparison blocks (n=42) during the previous academic year. Closed-ended items assessed beliefs about different aspects of Continuous Quality Improvement (CQI) project development and implementation (6 items). In addition, there were 5 short definition items to address knowledge. Finally, content analysis methods will be used to evaluate responses to the open-ended item which asked respondents to develop a project to improve patient care.
- Comparison Group: Alternate rotations and didn't receive intervention
Period: Overall Study
Arm/Group | PBL Curriculum Group | Comparison Group
Started | 50 | 42
Completed | 50 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No descriptive information was collected from subjects.
Groups:
- PBLI Curriculum Group: Received PBLI curriculum to evaluate and develop tools.
- Comparison Group: Didn't receive intervention
- Total: Total of all reporting groups
Arm/Group | PBLI Curriculum Group | Comparison Group | Total
Number analyzed (Participants) | 50 | 42 | 92
Age, Customized [Number; unit: participants] — Age was not collected
  participants | NA — Age was not collected as it was not relevant to the study focus. | NA — Age was not collected as it was not relevant to the study focus. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Number; unit: participants] — Gender was not collected
  participants | NA — Gender of participants was not relevant to study focus. | NA — Gender of participants was not relevant to study focus. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Beliefs About Ability to Implement a CQI Project
Description: Residents' belief about their ability to implement a CQI project was measured using a single efficacy item (values ranged from 1, strongly disagree, to 5, strongly agree). The item is from the Systems Quality Improvement Training and Assessment Tool. Differences (post minus pre) in this belief item were looked at with positive and higher difference values reflecting more positive change/increase in belief.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PBLI Curriculum Group: Received the intervention and used to evaluate and develop PBLI tools
Arm/Group | PBLI Curriculum Group | Comparison Group
Number analyzed (Participants) | 46 | 40
units on a scale | .80 (.81) | .28 (.93)
Statistical Analysis 1: Comparison: PBLI Curriculum Group vs Comparison Group; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Change in Knowledge Scores About Quality Improvement
Description: Residents' knowledge was assessed using the knowledge scale (e.g., describe change concept, how a cause-effect diagram is created, elements of the improvement model) from the SQI TAT and scores could range from 0 to 54 points. Difference scores were used based on total score of the scale with larger positive values indicating more increase in knowledge.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PBLI Curriclum Group: Received the intervention and evaluate and develop PBLI tools
- Comparison Group: Didn't receive the intervention.
Arm/Group | PBLI Curriclum Group | Comparison Group
Number analyzed (Participants) | 46 | 40
units on a scale | 4.39 (4.89) | 0.73 (2.51)
Statistical Analysis 1: Comparison: PBLI Curriclum Group vs Comparison Group; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- PBLI Curriculum Group: Received the intervention. To evaluate and develop PBLI tools.
Arm/Group | PBLI Curriculum Group | Comparison Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/42
Other Adverse Events (participants affected / at risk) | 0/50 | 0/42

LIMITATIONS AND CAVEATS:
While necessary limitations for initial assessment tool development, concerns will be addressed in the multi-site trial of the curriculum, including assessment of the training manual and codebooks that were developed during this project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No